CLINICAL TRIAL: NCT05766553
Title: Effects of Mindfulness Meditation in Virtual Reality on Craving and Smoking Cessation
Acronym: VIREAMIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A02004-39
Record Dates: First submitted 2023-01-18; First posted 2023-03-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Tobacco Use Disorder
Keywords: relapse; craving
MeSH Terms: conditions — Tobacco Use Disorder; Recurrence | interventions — Tobacco Use Cessation Devices; Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Patients in this arm will have 6 sessions of virtual reality in a pod (1 session per week).
  Patients will then have a visit at day 90 and day 180.
  Interventions: Other: Virtual reality pod
- Control group (Active Comparator): Patients in this arm will receive the gold standard of treatment for tobacco cessation (nicotine patches and chewing gum) from day 0 (inclusion visit) to day 90.
  Patients will then have a visit at day 90 and day 180.
  Interventions: Other: nicotine patches and chewing gum

INTERVENTIONS:
Other: Virtual reality pod — The first two sessions provide guided training in relaxation and mindfulness through immersion in a virtual forest environment for the first session, and in a virtual beach environment for the second. Sessions 3 and 4 present environments with addiction-related stimuli (Cues). The session 3 consists of a walk through the virtual street environment, buying a bottle of water from the store, and then ordering a coffee from a virtual bar. The session 4 takes place in a virtual party environment in an apartment: people smoke and drink alcohol in the living room, the session consists of sitting with them, then going to the kitchen to get a water bottle. Sessions 5 and 6 present stressful environments. Session 5 consists of a virtual parachute jump. The 6th session takes place in a virtual airplane environment, which will encounter turbulence.
  Arms: Interventional Group
Other: nicotine patches and chewing gum — Participants in this group will be prescribed a Gold Standard smoking cessation treatment with nicotine patches adapted to their consumption and 4mg nicotine chewing gum for a period of 3 months.
  Arms: Control group

SUMMARY:
Investigators seek to propose a non-drug therapeutic alternative, namely a mindfulness meditation protocol based on virtual reality training in order to induce progressive modifications of various indicators of craving.

The study hypothesis is that the practice of mindfulness meditation in a virtual reality environment reduces the craving induced by cues and stress and therefore ultimately smoking relapse.

The main objective of the protocol will be to demonstrate that mindfulness meditation can reduce long-term relapse (continuous cessation (> 30 days) of smoking cessation).

The participants will be randomized into two groups: the experimental group will perform six virtual reality sessions in a multisensory cabin at the rate of one session per week; the control group will be prescribed the gold standard treatment (nicotine patches and chewing gum).

Participants will be seen again at three and six months to assess whether or not there has been a smoking relapse.

ELIGIBILITY:
Inclusion Criteria:

* Any patient consuming 10 to 40 cigarettes per day
* Woman or man aged 18 to 75 inclusive
* Substance use disorder according to the DSM5 classification
* Benefit from social security or benefit from it through a third party in accordance with French law on research involving the human person
* Having signed the informed consent form after having received written information.

Exclusion Criteria:

* Disabling cognitive disorders
* Patient under 18 or over 75 years old.
* Patient with a psychological disorder or a psychiatric pathology requiring specialized follow-up
* Patient with addiction to another product.
* Cardiological pathologies that could compromise the participation of patients, detected by an ECG (only for patients who will be randomized in the experimental group).
* Advanced pulmonary, renal, and hepatic diseases, or any unstable and serious medical conditions that could compromise the patient's participation in the study, subject to the judgment of the doctor
* Pregnant or breastfeeding woman
* Simultaneous participation in another trial
* Employee of the investigator or of the clinical trial site
* Patients protected by law
* Patients who do not speak the French language
* People not covered by state health insurance
* Patients who in the opinion of the investigator are unable to complete the questionnaires
* Patient claustrophobic or anxious about using the cabin
* Patient allergic to a molecule present in nicotine substitutes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Relapse at 3 months | 3 months
  Relapse of patients by declaring their consumption at 3 months.
Relapse at 6 months | 6 months
  Relapse of patients by declaring their consumption at 6 months.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Cabinet Médical, Iteuil
  - Cabinet médical des Couronneries, Poitiers
  - Centre Hospitalier Henri Laborit, Poitiers